CLINICAL TRIAL: NCT01848912
Title: Temperature, Heart and Respiratory Rate Investigation Along With Variability Evaluation and Serum Biomarkers (THRRIVES)
Acronym: THRRIVES
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 20120564-01H
Record Dates: First submitted 2013-04-18; First posted 2013-05-08 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bone Marrow Transplant Patients
  Interventions: Device: Zephyr Biopatch Device

INTERVENTIONS:
Device: Zephyr Biopatch Device

SUMMARY:
The purpose of this study is to find a way of detecting infection earlier in patients receiving bone marrow transplant. This is accomplished by continuous individualized monitoring of heart rate, respiratory rate and temperature variability in this patient population. The investigators are collecting data to determine whether or not subtle differences in heart rate, respiratory rate and temperature will help physicians to detect infection earlier in order to begin faster treatment before a patient's condition deteriorates. Blood tests will also be performed to check for certain biomarkers that may indicate infection

DETAILED DESCRIPTION:
In this prospective observational study, patients receiving bone marrow transplant are selected for continuous monitoring of heart rate, respiratory and temperate variability. Data is collected as per standard practice using the Zephyr Biopatch device, a highly compact wireless monitor with two small gel electrodes, that is much more comfortable than previous belt/strap-based monitoring devices.

The patient is asked to wear the Zephyr Biopatch device for approximately 23 hours a day, beginning the day before he/she begins bone marrow transplant. The patient is asked to continue wearing the device for a period of up to 10 days or until he/she is no longer experiencing any fever. The Zephyr Biopatch device records heart rate, respiratory rate and temperature for calculation of heart rate variability (HRV), respiratory rate variability (RRV) and temperature variability (TV) using the Continuous Multiorgan Individualized Variability Analysis (CIMVATM) software engine. The variability outcomes will look at the presence, rapidity and severity of change in variability prior to the onset, diagnosis and treatment of infection. Bloodwork will also be performed to check for certain biomarkers that may indicate infection.

ELIGIBILITY:
Inclusion Criteria:

An expected prolonged period of neutropenia

* Completing bone marrow;
* Allogeneic and/or autologous transplants OR
* Induction chemotherapy

Exclusion Criteria:

* Inability to obtain written informed consent from patient or legally authorized representative
* Ongoing treatment for active infection (not prophylaxis)
* Preexisting severe cardiopulmonary disease (defined as an EF 40%, FEV 40%,or interstitial lung disease with pulmonary fibrosis)
* On betablockers or calcium channel blockers
* Preexisting arrhythmia
* Permanent pacemaker
* Inability to speak neither English nor French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an expected prolonged period of neutropenia completing bone marrow transplant (including both allogeneic and autologous) or induction chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2013-03; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Initiation or broadening of antibiotic for the purpose of treatment of infection | Patients are monitored for a period of up to 10 days or until their white blood cell count goes up, which could take an expected average of 20 days

SECONDARY OUTCOMES:
Admission to ICU with organ failure or hospital | Patients are monitored for a period of up to 10 days or until their white blood cell count goes up, which could take an expected average of 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bredeson, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute; Andrew Seely, MD, PhD, Study Director — Ottawa Hospital Research Institute; Bill Cameron, MD, FRCPC, Study Chair — Ottawa Hospital Research Institute; Tim Ramsay, MSc, PhD, Study Chair — Ottawa Hospital Research Institute; Lauralyn McIntyre, MD MSc, Study Chair — Ottawa Hospital Research Institute; Lothar Huebsch, MD, Study Chair — Ottawa Hospital Research Institute
Locations (1):
- Bone Marrow Transplant Clinic,The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided